CLINICAL TRIAL: NCT05159973
Title: Frequency of Serious Rhythmic Complications in Patients With Non-ST-segment Elevation Acute Coronary Syndrome
Brief Title: Patients With Non-ST-segment Elevation Acute Coronary Syndrome
Acronym: SCA
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8410
Record Dates: First submitted 2021-11-17; First posted 2021-12-16 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Myocardial Infarction
Keywords: Acute Coronary Syndrome; ACS; ST segment elevation; Myocardial infarction
MeSH Terms: conditions — Myocardial Infarction; Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
There are two types of acute coronary syndrome (ACS): ACS with persistent ST segment elevation (ACS ST +) and ACS without ST segment elevation (non-ST + ACS). The incidence of non-ST + ACS is increasing and currently accounts for the majority of myocardial infarction (MI) hospitalizations, while that of ST + ACS is declining. Complications of MI, which include rhythm and conduction disturbances, are mainly associated with ACS ST +. It is recognized that these complications can occur during non-ST + ACS, but with less frequency. This frequency is not clearly established, and has been the subject of few studies. Recent studies in this direction suggest that the frequency of rhythmic complications is low during non-ST + ACS. However, the data collected concerns inter-hospital transport.

The aim of the study is to estimate the frequency of occurrence of potentially fatal rhythmic complications in patients admitted to the emergency room and to the cardiology department for non-ST + ACS.

ELIGIBILITY:
Inclusion criteria:

* Adult patient (≥ 18 years old)
* Man or woman
* Patient admitted to the Emergency Department (SU) or to the Cardiology Department at the NHC between January 1, 2019 and December 31, 2020
* Patient whose main diagnosis retained at the end of hospitalization is a non-ST + ACS
* Patient who did not express his opposition to the reuse of his data for scientific research purposes.

Exclusion criteria:

* Subject having expressed opposition to participating in the study
* Subject under guardianship, curatorship or safeguard of justice

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patient whose main diagnosis retained at the end of hospitalization is a non-ST + ACS
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-09-21 (Actual); Study Completion 2022-09-21 (Actual)

PRIMARY OUTCOMES:
Evaluation of the frequency of occurrence of potentially fatal rhythmic complications in patients with non-ST segment elevation acute coronary syndrome | Files analysed retrospectively from January 01, 2019 to December 31, 2020 will be examined]

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien HARSCOAT, MD, Principal Investigator — Service des Urgences Médico-Chirurgicales Adultes - Hôpitaux Universitaires de Strasbourg
Locations (1):
- Service des Urgences Médico-Chirurgicales Adultes - Hôpitaux Universitaires de Strasbourg, Strasbourg, France